CLINICAL TRIAL: NCT00538772
Title: An Exploratory Correlative Study of Biomarkers in Patients With Metastatic Renal Cell Carcinoma Who Have Progressed After Sunitinib Therapy
Status: Withdrawn | Type: Observational
Sponsor: Kim Chi (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Kim Chi, Medical Oncologist, British Columbia Cancer Agency
Organization: British Columbia Cancer Agency (Other)
Other Study IDs: KNC-001; Biomarkers; Metastatic Renal Cell
Record Dates: First submitted 2007-09-28; First posted 2007-10-03 (Estimated); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Carcinoma, Renal Cell
Keywords: Metastatic Renal Cell Carcinoma; Biomarkers; Biomarkers in patients with Metastatic Renal Cell Carcinoma Who Have Progressed After Sunitinib Therapy
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Approx. 40ml of blood for correlative studies will be drawn at predetermined time points: baseline, after cycle 1, at time of treatment failure/discontinuation of protocol therapy.
  10 unstained slides from original patient specimen (nephrectomy specimens only) will be collected within 6 months after enrollment.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Biomarker
  Interventions: Other: Not applicable - blood tests/tissue specimen tests will be undertaken

INTERVENTIONS:
Other: Not applicable - blood tests/tissue specimen tests will be undertaken — Not applicable - blood tests/tissue specimen tests will be undertaken

SUMMARY:
Purpose:

The purpose of the correlative studies is to evaluate levels of serum factors of circulating VEGF and soluble VEGFR, circulating tumor cells and circulating endothelial cells assayed at baseline and over the course of initial treatment in order to explore relationships with baseline patient factors, measurable disease response and clinical progression.

Hypothesis soluble markers of angiogenic growth factors and receptors, and circulating endothelial and tumor cells can serve as markers for biologic activity of temsirolimus and/or sorafenib.

DETAILED DESCRIPTION:
It is recognized that the measurable disease RECIST criteria response rate with mTOR inhibition is likely to be low and that the benefit of such therapy will also include effects on disease stabilization. Disease stabilization is difficult to interpret in the phase II setting. Thus, it is desirable to develop biomarkers which will provide additional information on novel treatment effects and how they might relate to disease progression

ELIGIBILITY:
Inclusion Criteria:

* All patients enrolled from Canadian centres for the Wyeth Pharmaceuticals sponsored multicenter, open-label phase III study evaluating second line therapy with either temsirolimus or sorafenib in patients progressing after sunitinib therapy, are eligible for this correlative studies protocol.
* Patients must provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects from Canadian centres who have agreed to participate in the trial entitled "A randomized trial of Temsirolimus and Sorafenib as second line therapy in patients with advanced renal cell carcinoma who have failed first line Sunitinib therapy" will be approached to participate in this Exploratory Biomarker study
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-07; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
This is an exploratory study. Correlations between biomarkers and baseline factors and treatment outcomes will be made | Not available as study withdrawn on November 2010

CONTACTS AND LOCATIONS:
Overall Officials: Christian Kollmannsberger, MD, Principal Investigator — BC Cancer Agency- Vancouver
Locations (3):
- Canada (3):
  - BC Cancer Agency - Centre for Southern Interior, Kelowna, British Columbia
  - BC Cancer Agency - Vancouver, Vancouver, British Columbia
  - BC Cancer Agency - Vancouver Island, Victoria, British Columbia